CLINICAL TRIAL: NCT01857219
Title: A Brain Imaging Study of Tai Chi on Fibromyalgia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2012P002574
Record Dates: First submitted 2012-12-06; First posted 2013-05-20 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Fibromyalgia
Keywords: fMRI
MeSH Terms: conditions — Fibromyalgia | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Role of Tai Chi in Fibromyalgia (Experimental): Each Tai Chi session will last 60 minutes and will continue twice a week for 12 weeks. Our instructors, who have extensive experience conducting Tai Chi training programs, will follow the standardized Tai Chi protocol. We will also provide the participants with printed materials on FM and the Tai Chi Mind-Body program, including Tai Chi principles, practicing techniques, and safety precautions for participants with FM.
  In the first session, the Tai Chi instructors will explain exercise theory and procedures of Tai Chi. For the remaining sessions, the subjects will practice Tai Chi under the instruction of one of the Tai Chi instructors. Every session will include the following components: (1) warm-up and self-massage and a review of Tai Chi principles; (2) Tai Chi movement; (3) breathing techniques; (4) relaxation. Each component of the program derives from classical Yang style Tai Chi 108 posture.30
  Interventions: Behavioral: Tai chi

INTERVENTIONS:
Behavioral: Tai chi

SUMMARY:
To accomplish our Specific Aims, we propose to conduct a two-session fMRI experiment in up to 30 patients with fibromyalgia (FM) and up to 30 healthy controls. All subjects will be invited to complete the second, identical fMRI session about 3 months following completion of the first session. Fibromyalgia subjects will complete their scans before and after a 12-week Tai Chi intervention in collaboration with Tufts Medical Center.

ELIGIBILITY:
Criteria for fibromyalgia patients.

Inclusion Criteria:

* Volunteers 18-50 years of age.
* Fibromyalgia for at least the past 3 months, as determined by the referring physician.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Specific causes of pain (e.g., cancer, fractures, spinal stenosis, infections)
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome.
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.

Criteria for healthy adults.

Inclusion Criteria:

* Volunteers 18-50 years of age.
* At least a 10th grade English-reading level; English can be a second language provided that the patients feel they understand all the questions used in the assessment measures.

Exclusion Criteria:

* Chronic and acute pain (ex. Fibromyalgia).
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome.
* Presence of any contraindications to fMRI scanning. For example: cardiac pacemaker, metal implants, fear of closed spaces, pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-11 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Arterial spin labeling (ASL) before and after Tai Chi intervention. | 12 weeks
  A method to assess cerebral blood flow change (at rest) through functional magnetic in resonance imaging in response to Tai Chi intervention.

SECONDARY OUTCOMES:
Resting-state BOLD fMRI before and after Tai Chi intervention. | 12 weeks
  A method to measure spontaneous brain activity fluctuations through functional magnetic resonance imaging in response to Tai Chi intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Kong, MD, MPH, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States